CLINICAL TRIAL: NCT00505492
Title: A Phase II Study of Adjuvant Postoperative Radiation With Cisplatin Followed by Carboplatin/Paclitaxel Chemotherapy Following Total Abdominal Hysterectomy/Bilateral Salpino-Oophorectomy (TAH/BSO) for Patients With Stage I, II and IIIa Malignant Mixed Mesodermal Tumor (MMMT) of the Uterus.
Brief Title: Malignant Mixed Mesodermal Tumor (MMMT) - Early Stage With Postoperative XRT/Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-535
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Uterine Neoplasms
Keywords: Malignant Mixed Mesodermal Tumor; MMMT; Uterine Neoplasms; Radiation Therapy; Paclitaxel; Carboplatin; Cisplatin; Taxol
MeSH Terms: conditions — Uterine Neoplasms; Carcinosarcoma | interventions — Carboplatin; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation + Chemotherapy (Experimental): Radiation with weekly Cisplatin 40 mg/m^2 intravenously (IV) Followed by Carboplatin (AUC 5 IV)/Paclitaxel (135 mg/m^2 IV) Chemotherapy every 28 days
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — AUC 5 by vein once every 28 Days
  Other Names: paraplatin
Drug: Cisplatin — 40 mg/m^2 by vein (IV) Weekly Over 4 Hours
  Other Names: Platinol-AQ; Platinol; CDDP
Drug: Paclitaxel — 135 mg/m^2 by vein (IV) Once Every 28 Days
  Other Names: Taxol

SUMMARY:
Primary Objectives:

1. To test whether the addition of chemotherapy to radiotherapy improves the progression-free survival for patients with stage I, II and IIIa malignant mixed mesodermal tumor (MMMT) of the uterus.
2. To determine the acute and late toxicity profiles associated with this treatment regimen.
3. To describe the effect of this treatment regimen on the patient's quality of life.

DETAILED DESCRIPTION:
Patients in this study will have an operation to remove their uterus, tubes, and ovaries with biopsies of the omentum and lymph nodes before entering this study.

Before treatment starts, patients will have a chest x-ray, computed tomography (CT) scan, blood tests, and a physical exam. Patients who have a history of hearing loss will have a hearing test.

Within 8 weeks after surgery, patients will receive 5 weeks of combination radiation therapy and cisplatin chemotherapy. Radiation and cisplatin will be given on Day 1 or day 2 of each week followed by 4 days of radiation alone. An additional dose of radiation, directed at the surface of the vagina, will be given either during the last week (Week 5) of treatment or after the radiation and cisplatin chemotherapy is finished.

Three to five weeks after radiation therapy and cisplatin chemotherapy is finished, patients will receive additional chemotherapy. Carboplatin and paclitaxel will be given every 28 days for 4 cycles. All chemotherapy is given into the vein through a catheter (tube).

Patients will be taken off study if their disease gets worse or intolerable side effects occur. Patients will be seen one month after the last cycle of chemotherapy, then every 3-4 months from then on for 2 years. At each visit, patients will have blood tests and a physical exam. Computed tomography (CT) scans will be ordered only if it is suspected that the disease has come back. All patients will be followed for a maximum of 2 years after their therapy is completed.

This is an investigational study. Cisplatin, Carboplatin and Paclitaxel are FDA approved and commercially available. A total of 49 patients will take part in this study. Up to 25 patients may be enrolled at M. D. Anderson Cancer Center in Houston, up to 12 patients will be enrolled at MD Anderson Cancer Center, Orlando, and up to 12 patients will be enrolled at the University of Texas Medical Branch in Galveston.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed malignant mixed mesodermal (MMMT) confined to the pelvis (Stage IB, IC, IIA, IIB, IIIA).
* Patients who have undergone a total abdominal hysterectomy, vaginal hysterectomy or laparoscopic assisted vaginal hysterectomy and a bilateral salpino-oophorectomy (with minimal surgical staging, including omental biopsy and lymph node sampling) within 8 weeks of study entry.
* No known metastatic extrauterine metastases, no known gross residual disease or distant metastases.
* Women of any racial or ethnic group are eligible.
* Zubrod performance status of </= 2.
* Adequate bone marrow, renal and hepatic function: Hgb > 10 gm/dl, ANC >1.5/mm3, Platelets > 100,000/mcl, Creatinine < 1.5 mg/%, Bilirubin < 2.5 mg/dl, SGPT < 2* ULN, BUN < 1.5* ULN.
* No prior chemotherapy or radiation therapy for this diagnosis.
* Estimated life expectancy of 12 weeks or greater.
* Must sign an institutionally approved informed consent.

Exclusion Criteria:

* Previously treated malignant mixed mesodermal (MMMT) with either chemotherapy or radiotherapy (XRT)/
* Patients with gross residual disease, suspected extrapelvic or extrauterine disease or distant metastatic disease (Stage IIIB, IIIC or IV).
* History of other malignancy, with the exception of non-melanomatous skin cancer, unless in complete remission and off all therapy for that disease for a minimum of 5 years.
* Patients with a Zubrod performance status of 3 or greater.
* Patients with an active systemic infection.
* Patients with a serious intercurrent medical illness.
* Patients with a recent (within 6 months) history of cardiac dysrhythmia, congestive heart failure, unstable angina or myocardial infarction.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2002-02; Primary Completion 2006-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 7 Years
  Survival defined as observed length of life from study entry until death or, for living patients, date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Lois M. Ramondetta, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - UT MD Anderson Cancer Center, Houston, Texas
  - University of Washington School of Medicine, Seattle, Washington

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org